CLINICAL TRIAL: NCT05381103
Title: PSMA-PET to Guide Prostatectomy: A Randomized Trial
Brief Title: PSMA-PET to Guide Prostatectomy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Five Eleven Pharma, Inc. (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IU_CLN02_EPE
Record Dates: First submitted 2022-04-29; First posted 2022-05-19 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PSMA-PET and SOC MRI prior to surgery (Experimental)
  Interventions: Diagnostic Test: PSMA-PET and SOC MRI
- SOC MRI prior to surgery (Active Comparator)
  Interventions: Diagnostic Test: SOC MRI

INTERVENTIONS:
Diagnostic Test: PSMA-PET and SOC MRI — 60 min continuous acquisition of PET data after 3-6 mCI injection of [68Ga]P16-093 followed by contrast-CT
  Arms: PSMA-PET and SOC MRI prior to surgery
Diagnostic Test: SOC MRI — Standard of care MRI
  Arms: SOC MRI prior to surgery

SUMMARY:
In this study, 196 patients will be randomized 1:1 to either having only the standard of care MRI prior to surgery versus having the standard of care MRI and the PSMA PET scan. PET (and MRI) findings will be validated against whole mount pathology. Pre-surgical imaging findings will also be evaluated in the context of affecting subsequent surgical plans and impacting actual patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Significant prostate cancer:

   Gleason 3+4 ≥1 core with pattern 4 ≥20%

   Gleason 3+4 ≥1 core with ≥50% total involvement of core OR ≥3 cores of Gleason 3+4 OR

   NCCN unfavorable intermediate risk OR

   Any Gleason 4+3, 4+4, 4+5, 5+4, or 5+5 AND
2. Baseline sexual function (IIEF-EF > 17): No erectile dysfunction OR mild-to- moderate erectile dysfunction (International Index of Erectile Function Domain ≥ 17) AND
3. The patient desires to maintain erections following treatment
4. Planned to undergo a standard of care MRI or recently completed standard of care MRI within 6 months of scheduled date of surgery. Note: For subjects whose SOC MRI is not within 6 months or not 3Tesla, they may be enrolled in the study and the MRI will be repeated as a research study. The research MRI will not be billed to the subject's insurance, but will be scheduled at IU ORI, at no cost to study participant.
5. Planned Prostatectomy candidate per treating oncologist with prostatectomy planned within 90 days of consent.

Exclusion Criteria:

1. Participation in another investigational trial involving research exposure to ionizing radiation concurrently or within 30 days.
2. Does not meet safety criteria for MRI scan (e.g. metal implant that is not allowed, since MRI is required for comparison).
3. Significant acute or chronic medical, neurologic, or illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-EF sub scale score | 1 month
  International Index Erectile Function-Erectile Function sub scale score. Maximum score is 30 with higher score indicating better outcomes.
IIEF-EF sub scale score | 3 months
  International Index Erectile Function-Erectile Function sub scale score. Maximum score is 30 with higher score indicating better outcomes.
IIEF-EF sub scale score | 6 months
  International Index Erectile Function-Erectile Function sub scale score. Maximum score is 30 with higher score indicating better outcomes.
IIEF-EF sub scale score | 12 months
  International Index Erectile Function-Erectile Function sub scale score. Maximum score is 30 with higher score indicating better outcomes.
IIEF-EF sub scale score | 18 months
  International Index Erectile Function-Erectile Function sub scale score. Maximum score is 30 with higher score indicating better outcomes.

SECONDARY OUTCOMES:
Change in treatment plan | 1 month
  Proportion of patients whose treatment plan would be changed by PSMA-PET. Treatment changes are defined as any change in surgical resection plan that affects one of 4 critical regions for quality of life
Ratio of positive surgical margins to nerve bundles spared | 1 month
EPE detection | 1 month
  Sensitivity/Specificity for extra-prostatic extension of cancer at the nerve bundles
Incontinence bother | 18 months
  Expanded Prostate Cancer Index Composite (EPIC-26) questions 1-2
Incontinence: using 0-1 pads per day | 18 months
  Expanded Prostate Cancer Index Composite (EPIC-26) question 3
Urgency/frequency | 18 months
  Expanded Prostate Cancer Index Composite (EPIC-26) questions 4-5
Erectile dysfunction: ability to achieve erection sufficient for penetration | 18 months
  IIEF question 3
Overall mental and physical health | 18 months
  Short Form quality of life questionnaire (SF-36)
Surgical margins | 1 month
  postive surgical margin rates

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Bahler, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Goodman Hall, Indiana Institute for Biomedical Imaging Sciences, Indiana University School of Medicine, Indianapolis, Indiana, United States